CLINICAL TRIAL: NCT03510182
Title: Transcranial Direct Current Stimulation (tDCS) and Intensive Therapy in Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Carol Persad, Associate Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00108213
Record Dates: First submitted 2018-04-05; First posted 2018-04-27 (Actual); Results first posted 2021-09-20 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-08

CONDITIONS: Aphasia
MeSH Terms: conditions — Aphasia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: All eligible participants with aphasia will receive the tDCS
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- transcranial Direct Current Stimulation (Experimental): tDCS will be given to all qualified patients with aphasia.
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation

SUMMARY:
Intensive therapy for aphasia has been demonstrated to improve language functioning after stroke or other neurological injury. However, recovery is generally not complete and new therapies are needed to improve outcomes. Transcranial direct current stimulation (tDCS) has been shown to improve outcomes with motor therapy after stroke. This study will examine the feasibility of using tDCS with intensive language therapy as a way of enhancing language outcomes in aphasia

DETAILED DESCRIPTION:
Intensive therapy for aphasia has been demonstrated to improve language functioning after stroke or other neurological injury. However, recovery is generally not complete and new therapies are needed to improve outcomes. Transcranial direct current stimulation (tDCS) has been shown to improve outcomes with motor therapy after stroke. This study will examine the feasibility of using tDCS supplementing clinically determined intensive language therapy as a way of enhancing language outcomes in aphasia. Eligible clients enrolled in the University of Michigan Aphasia Program (UMAP) will be invited to participate in the study. Clients will receive 20 minutes of tDCS every day along with their usual treatment protocol. Pre and post testing will be completed to assess for improvement in language functioning. This is a feasibility and proof of concept study to determine if a randomized control trial should be pursued

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of aphasia
* Enrolled in intensive therapy program at the University of Michigan Aphasia Program.
* Ability to understand and give consent to treatment.

Exclusion Criteria:

* No metal implants or surgical devices
* History of seizures
* History of significant cognitive or psychiatric disturbance
* Participant cannot be pregnant at the time of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol Persad, PhD, Principal Investigator — University of Michigan
Locations (1):
- University Center for Language and Literacy, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Transcranial Direct Current Stimulation: tDCS will be given to all qualified patients with aphasia.
  transcranial direct current stimulation
Period: Overall Study
Arm/Group | Transcranial Direct Current Stimulation
Started | 25
Completed | 23
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Boston Naming Test [Mean (Standard Deviation); unit: units on a scale] — This test assesses confrontational naming ability to 60 line drawings. Scores range from 0-60 with higher scores representing better performance.
  units on a scale | 5.94 (5.97)
Controlled Oral Word Fluency [Mean (Standard Deviation); unit: number of words] — This test assesses the number of words that can be generated in one minute that begin with certain letters. The total number of words generated for three letters is derived. Higher scores represent better performance.
  number of words | 14.74 (10.27)

OUTCOME MEASURES:

1. Primary Outcome: Change in Controlled Oral Word Fluency
Description: This test assesses the number of words that can be generated in one minute that begin with certain letters. The total number of words generated for three letters is derived. Higher scores represent better performance. Changes in word fluency were calculated as follows: number of words generated post tDCS minus number of words generated pre tDCS
Time Frame: baseline and 4 weeks
Population: 23 of the participants completed the study
Measure: Mean (Standard Deviation); unit: number of words
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 23
number of words | 3.1 (4.89)

2. Primary Outcome: Change in Boston Naming Score
Description: This test assesses confrontational naming ability to 60 line drawings. Scores range from 0-60 with higher scores representing better performance. Outcome was derived as followed : Picture naming score post tDCS minus picture naming score pre tDCS
Time Frame: baseline and 4 weeks
Population: 23 of the 25 subjects completed the study and their data are analyzed here
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 23
score | 1.25 (3.96)

3. Secondary Outcome: Change in Western Aphasia Quotient Score
Description: severity of aphasia is measured by the Western Aphasia Battery Revised. The Aphasia Quotient (AQ) score ranges from 0-100, with 100 being a perfect score. Change in the AQ was derived as follows : AQ post tDCS minus AQ pre tDCS
Time Frame: baseline and 4 weeks
Population: 23 subjects completed the study and their data were analyzed
Measure: Mean (Standard Deviation); unit: aphasia quotient score
Arm/Group | Transcranial Direct Current Stimulation
Number analyzed (Participants) | 23
aphasia quotient score | 8.57 (6.37)

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Transcranial Direct Current Stimulation
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-10): https://cdn.clinicaltrials.gov/large-docs/82/NCT03510182/Prot_SAP_000.pdf